CLINICAL TRIAL: NCT01731392
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Effect of Milk-based Formulas on Infections and Immune Functions in Healthy Children
Brief Title: Children Immune Functions(2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10.50.NRC
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Diarrhea; Upper Respiratory Infections
Keywords: Diarrhea; Children; Lactobacilli
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk with Bifidobacteria (Experimental): duration of the treatment is 5 months
  Interventions: Dietary Supplement: Milk with Bifidobacteria
- Milk with non replicating lactobacilli (Active Comparator): duration of the treatment is 5 months
  Interventions: Dietary Supplement: Milk with non replicating lactobacilli
- Semi skimmed milk (Placebo Comparator): duration of the treatment is 5 months
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Milk with Bifidobacteria — A total of 36g (4 spoons) of powder milk per serving are diluted in 220 ml of water. Two servings per day are consumed orally, corresponding to 72g per day.
  Arms: Milk with Bifidobacteria
Dietary Supplement: Milk with non replicating lactobacilli — A total of 36g (4 spoons) of powder milk per serving are diluted in 220 ml of water. Two servings per day are consumed orally, corresponding to 72g per day.
  Arms: Milk with non replicating lactobacilli
Dietary Supplement: placebo — A total of 36g (4 spoons) of powder milk per serving are diluted in 220 ml of water. Two servings per day are consumed orally, corresponding to 72g per day.
  Arms: Semi skimmed milk

SUMMARY:
To investigate the effect of milk-based formulas on infections and immune functions in healthy children.

DETAILED DESCRIPTION:
Particular attention was paid to the role played by nutrition in supporting the gut ecosystem, balancing microbiota and promoting health status. In that respect, the beneficial effects of probiotics were demonstrated for different infectious diseases, GII and URI.

The beneficial effect of probiotics for treatment of symptomatic diarrhea was clearly documented.

ELIGIBILITY:
Inclusion Criteria:

* Parents written and signed informed consent for participation in the study.
* Healthy children aged 1 to 3 years that are no more breastfed.
* Go to a selected nursery and / or pediatrician.
* Parents must have a phone at home or a cellular phone to call the paediatrician.
* No consumption of commercial products containing probiotics or prebiotics during the 3 weeks before and during the study period.
* Parents are able to give their children, twice daily, 2 milk servings on a 5 months period.
* Children not being intensive consumers of regular yoghurts

Exclusion Criteria:

* Rotavirus and flu vaccines administration within the last 3 months prior to V1 (baseline visit).
* Used antibiotics within the last 30 days prior to V1 (baseline visit).
* Congenital or chronic disease.
* Any kind of immunodeficiency or allergy, milk protein allergy or lactose intolerance.
* Significant illness within the two weeks prior to start of the study or any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 604 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Days with diarrhea | during the 5 months of follow up

SECONDARY OUTCOMES:
Number of episodes of Upper Respiratory Infections | 5 months
Duration of episodes of Upper Respiratory Infections | 5 months
Severity of episodes of Upper Respiratory Infections | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Saptawati Bardosono, MSc, Principal Investigator — Nutrition Department, Faculty of Medicine,
Locations (1):
- Dept. Nutrition, Faculty of Medicine University of Indonesia, Jakarta, Indonesia